CLINICAL TRIAL: NCT06728982
Title: Metformin Enhances Pathological Complete Response in Non-Diabetic Rectal Cancer Patients Undergoing Neoadjuvant Chemoradiotherapy: A Randomized Controlled Trial
Brief Title: Impact Of Metformin In Rectal Cancer Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Omar Mohamed Awad, Teaching Assistant, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Metformin In Rectal Cancer
Record Dates: First submitted 2024-11-29; First posted 2024-12-11 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-05

CONDITIONS: Rectal Cancer Patients
Keywords: metformin; complete pathological response; rectal patient; neoadjuvant chemoradiotherapy
MeSH Terms: conditions — Pathologic Complete Response | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups:
  Group A: Patients will receive standard chemoradiotherapy(CRT).
  Group B: Patients will self-administer 1000mg of metformin twice daily by mouth:
  1. beginning 1-2 weeks before standard CRT.
  2. during standard CRT.
  3. until 30 days after the end of standard CRT.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (No Intervention): Patients will receive standard chemoradiotherapy(CRT)
- Group B (Metformin) (Active Comparator): Patients will self-administer 1000mg of metformin twice daily by mouth:
  1. beginning 1-2 weeks before standard CRT.
  2. during standard CRT.
  3. until 30 days after the end of standard CRT.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 1000mg of metformin twice daily by mouth
  Arms: Group B (Metformin)

SUMMARY:
Design: Prospective, randomized controlled clinical trial Setting: at Minia University Hospital and Minia Oncology Institute. Condition: Colorectal cancer.

To be eligible for participation, patients must meet the following criteria:

1. Histologically confirmed diagnosis of rectal adenocarcinoma.
2. Age starting from 18 and older.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
4. Adequate organ function (renal, hepatic, and hematological)
5. Signed informed consent.

Patients will be randomized into two groups:

Group A: Patients will receive standard chemoradiotherapy(CRT).

Group B: Patients will self-administer 1000mg of metformin twice daily by mouth:

1. beginning 1-2 weeks before standard CRT.
2. during standard CRT.
3. until 30 days after the end of standard CRT.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of rectal adenocarcinoma.
2. Age starting from 18 and older.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
4. Adequate organ function (renal, hepatic, and hematological)
5. Signed informed consent.

Exclusion Criteria:

1. Metastatic disease.
2. Contraindications to metformin.
3. Significant comorbidities or medical conditions that may interfere with study participation. (D.M, PCO,..)
4. eGFR less than 30 mL/min.
5. Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) rate | 6 months
  The Main outcome is to assess the use of metformin to improve pathological complete response (pCR) rates among non-diabetic participants undergoing standard neoadjuvant CRT for rectal cancer.
  The primary outcome will be measured by the pathological complete response rate after completion of the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Omar M Awad, Bsc, Principal Investigator — Deraya University; Fatma M Mady, professor, Study Chair — Minia University; Mona A Saber, PhD, Study Director — Minia University
Locations (2):
- Egypt (2):
  - Minia Oncology Center, Minya, Egypt
  - Minia University Hospital, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No